CLINICAL TRIAL: NCT02445170
Title: Heath-related Quality of Life of Diabetic Transmetatarsal Amputees and Below-knee Prosthetic Users
Status: Withdrawn | Type: Observational
Why Stopped: The study is not eligible at present.
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jussi Repo, Researcher, Helsinki University Central Hospital
Other Study IDs: 364/13/03/02/2014/8
Record Dates: First submitted 2015-05-08; First posted 2015-05-15 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Amputees; Diabetes Complications
Keywords: Diabetes; amputation; below-knee; transmetatarsal; [M01.150.100]; [C19.246.099]
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus | interventions — Amputation, Surgical

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Below-knee amputees: The present group consists of diabetic below-knee prosthetic user
  Interventions: Procedure: Amputation
- Transmetatarsal amputees: The present group consists of diabetic transmetatarsal amputees
  Interventions: Procedure: Amputation

INTERVENTIONS:
Procedure: Amputation — Transmetatarsal or below-knee amputation

SUMMARY:
The present study assesses the health-related quality of life of diabetic transmetatarstal and below-knee prosthetic user. The study design is cross-sectional with a retrospective review of patient hospital records and an assessment with patient-reported outcome measure.

DETAILED DESCRIPTION:
The present study aims to recruit 100 diabetic transmetatarsal and below-knee prosthetic user to assess the health-related quality of life (HRQoL) between these two patient groups. The 15D HRQoL instrument is applied. An additional comparison with the age-standardized Finnish general population will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes
* Transmetatarsal amputation
* Below-knee prosthetic user
* 2-5 years from surgery

Exclusion Criteria:

* No diabetes
* Other than transmetatarsal or below-knee amputation
* Below-knee amputation but not a below-knee prosthetic user
* Less than 2 years from the amputation
* Over 5 years from amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients who underwent transmetatarsal amputaion or below-knee prosthetic users in a time frame of 2-5 years from the amputation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life measured by the HRQoL score | 2-5 years

SECONDARY OUTCOMES:
The 15D health-related quality of life instrument | 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Erkki J Tukiainen, professor, Study Director — Helsinki University Hospital and Helsinki University
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland